CLINICAL TRIAL: NCT06723639
Title: Effects of Restoring Achilles Tendon Anatomy After a Rupture: A Randomized Controlled Trial
Brief Title: Restoring Anatomy of Ruptured Achilles Tendon
Acronym: RATAR
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Bispebjerg Hospital (Other)
Collaborators: Copenhagen University Hospital, Hvidovre (Other); Sahlgrenska University Hospital (Other)
Responsible Party: Principal Investigator, Rikke Høffner, Post doc, PhD, PT, Bispebjerg Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: H-24041516
Record Dates: First submitted 2024-12-04; First posted 2024-12-09 (Actual); Last update posted 2025-04-15 (Actual); Status verified 2024-11

CONDITIONS: Achilles Tendon Rupture
Keywords: Achilles tendon rupture; MRI; Surgery; Restore anatomy; Heel-rise test; Rehabilitation
MeSH Terms: interventions — Wound Healing; Sutures; Surgical Procedures, Operative; Conservative Treatment

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- NEWSUR (Experimental): Participants in this group will receive a new two-layer surgical technique followed by a detailed rehabilitation regime.
  Interventions: Procedure: A new two-layer surgical technique
- CONSER (Other): Participants in this group will receive standard non-surgical treatment followed by a detailed rehabilitation regime.
  Interventions: Other: Standard non-surgical treatment

INTERVENTIONS:
Procedure: A new two-layer surgical technique — A new double row suturing technique attempting to restore the length of the distinct soleus and gastrocnemius portions of the Achilles tendon.
  Other Names: Repair; Sutur; Operation
  Arms: NEWSUR
Other: Standard non-surgical treatment — Standard non-surgical treatment
  Other Names: Standard; Conservative; No surgery
  Arms: CONSER

SUMMARY:
The goal of this clinical trial is to investigate a new surgical approach to restore the anatomy of a ruptured Achilles tendon. We will use a new two-layer technique followed by rehabilitation and find out how it influence the patients clinical outcome, muscle and tendon structure, and function after one year and compare with a standard non-surgical approach followed by rehabilitation. Participants will be randomized to 1) NEWSUR: A new two-layer surgical technique followed by rehabilitation regime or 2) CONSER: A standard non-surgical treatment followed by rehabilitation .

We hypothesize that restoring the anatomy of the ruptured mid-substance Achilles tendon using a new two-layer surgery technique followed by rehabilitation will yield a more favorable patient reported outcome (ATRS) one year after rupture compared to standard non-surgical treatment followed by rehabilitation.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with a complete mid-substance Achilles tendon rupture based on clinical exam, including Thompson/Matles test, by an experienced physician.
* Presented within 14 days from injury.
* Understands and reads Danish.
* No contraindications for MRI.

Exclusion Criteria:

* Smoking
* Diabetes
* Other injuries affecting their lower limb function.
* Contralateral Achilles tendon rupture.
* Re-rupture.
* Anticoagulation treatment.
* Inability to follow rehabilitation or complete follow-up tests.
* Immunosuppressive treatment, including systemic corticosteroid treatment.
* Pregnant

Ages: 18 Years to 67 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-02-28 (Actual); Primary Completion 2027-07-01 (Estimated); Study Completion 2027-07-01 (Estimated)

PRIMARY OUTCOMES:
The Achilles tendon Total rupture score (ATRS) | At 1 year
  The Achilles tendon Total rupture score (ATRS) will be used. The ATRS is a patient-reported instrument with high reliability, validity, and sensitivity for measuring the outcome related to symptoms and physical activity after treatment in patients with a total Achilles tendon rupture. The scale is from 0-100. A score of 100 points indicates full function and no pain with lower scores indicating reduced function.

SECONDARY OUTCOMES:
Hourly sporting activity | 1 year
  Data on activity level of sporting activities (h/week), if patients return to the same sport, and if patients return to the same job as prior to the injury will be obtained.
Patient satisfaction | 1 year
  Patient satisfaction regarding activities of daily living and sport participation will be evaluated using a 5-point Likert scale for satisfaction. With responses ranging from 1 (strongly dissatisfied) to 5 (strongly satisfied).
Tampa Scale of Kinesiophobia | 26 weeks & 1 year
  Increased fear of movement can be a sequala after an Achilles tendon rupture. The Danish (and swedish in Sweden) version of the Tampa Scale of Kinesiophobia (TSK-11) will be used to assess fear of movement. The TSK-11 is scored on a 4-point Likert scale, with responses ranging from 1 (strongly disagree) to 4 (strongly agree). The lowest possible score, 11, denotes negligible or nonexistent kinesiophobia. The highest possible score, 44, denotes a severe fear of experiencing pain while moving.
Heel-rise test | 26 weeks & 1 year
  Heel-rise muscle function (height) and repetitions will be evaluated using a standardized heel-rise test.
Ultrasonography | 1 year
  Muscle fascicle length, pennation angle and thickness of the medial gastrocnemius muscle will be measured with B-mode ultrasonography. Power doppler flow in the Achilles tendon will be recorded in the area with the highest visible Power Doppler activity.
Magnetic resonance imaging (MRI) | 1 year
  A 3D MRI of both Achilles tendons will be obtained. An axial 6-point DIXON sequence will also be applied to assess free fat fraction of the muscles.The uninjured side will serve as an internal control for all measures.
Plantarflexion muscle strength | 1 year
  Maximal isometric plantar flexion muscle strength will be measured in 10-degree increments from 10 degrees of dorsiflexion to 20 degrees of plantarflexion with the knee in extension (soleus + gastrocnemius) and in flexion (primarily soleus) while seated (Biodex Multi-joint System 4 Pro, Biodex Medical Systems, USA)
Vertical jump performance | 1 year
  For the countermovement jump, participants are instructed to stand on one leg with their arms folded across their chest, perform a maximal vertical jump, and aim to land in the same spot on the force plate. For the drop jump, participants stand on one leg with their arms folded across their chest on a 20cm box. They then jump down onto the force plate and, upon landing, perform a maximal vertical jump. Each participant will complete three repetitions on each leg for both tasks. For the hopping task, participants stand on one leg with their arms at their sides, as if jumping rope. They performed 25 rhythmic jumps at a self-selected pace, trying to remain in the same spot. Each participant completed two repetitions of the hopping task on each leg
Ankle joint range of motion (ATRA) | 26 weeks & 1 year
  The passive ankle joint range of motion will be assessed as the Achilles tendon resting angle (ATRA) with the subject lying prone with the knee in full extension (ATRAext) and with the knee in 90 degrees of flexion (ATRAflex) bilaterally using a standard goniometer as previously described. The uninjured side will serve as an internal control.
Knee to wall test | 26 weeks & 1 year
  Ankle dorsiflexion range of motion will be measured with the knee extended and knee flexed positions of the weight bearing lunge test bilaterally.

CONTACTS AND LOCATIONS:
Locations (3):
- Denmark (2):
  - , Copenhagen University Hospital Bispebjerg-Frederiksberg Hospital, Copenhagen, Denmark., Copenhagen, Capital
  - Copenhagen University Hospital, Amager-Hvidovre, Copenhagen, Capital
- Sahlgrenska University Hospital, Gothenburg, Sweden

IPD SHARING:
Plan to Share IPD: Undecided